CLINICAL TRIAL: NCT00630513
Title: A Prospective, Double-blind, Multi Center, Randomized Clinical Study to Compare the Efficacy and Safety of Ertapenem 3 Days Versus Ampicillin-Sulbactam 3 Days in the Treatment of Localized Community Acquired Intra-abdominal Infection (IAI). (T.E.A. Study Three Days Ertapenem vs Three Days Ampicillin- Sulbactam)
Brief Title: T.E.A. Study Three Days Ertapenem Versus Three Days Ampicillin- Sulbactam
Acronym: TEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Dr. Fausto Catena MD PhD, University of Bologna - St Orsola-Malpighi University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T.E.A. Study
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2008-09

CONDITIONS: Intra-Abdominal Infection
Keywords: localized community acquired intra-abdominal infection (IAI); antibiotics; localized peritonitis; ertapenem
MeSH Terms: conditions — Intraabdominal Infections | interventions — Ertapenem; sultamicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- E (Experimental): 3 days regimen with Ertapenem
  Interventions: Drug: Ertapenem
- AS (Active Comparator): 3 days treatment with Ampicillin-Sulbactam
  Interventions: Drug: Ampicillin-Sulbactam

INTERVENTIONS:
Drug: Ertapenem — 3 days regimen with Ertapenem (1 g/day i.v.)
  Arms: E
Drug: Ampicillin-Sulbactam — 3 days treatment with Ampicillin-Sulbactam (AS 3g x 3/ day i.v.)
  Arms: AS

SUMMARY:
The aim of the study was to compare the activity (efficacy and safety) of Ertapenem administered according to a short treatment for three days versus a short treatment for three days with AS in patients with an community acquired IAI of mild to moderate severity.

DETAILED DESCRIPTION:
The study project is a prospective, randomized controlled investigation. The study will be performed in the Department of Transplant, General and Emergency Surgery of St Orsola-Malpighi University Hospital (Bologna, Italy), a large teaching institution, with the participation of all surgeons who accept to be involved in.

The study is designed and conducted in compliance with the principles of Good Clinical Practice regulations.

The tolerability and efficacy of a 3 days treatment with Ampicillin- Sulbactam (AS 3g x 3/ day i.v.) is compared a 3 days regimen with Ertapenem (1 g/day i.v.). in patients with localized peritonitis with a blinded evaluation of efficacy end points. Evaluation of cure or failure is blinded by use of designated third party individuals who are unaware of the treatment assigned to the patients.

ELIGIBILITY:
Inclusion Criteria:

Adult patients ( > 18 years) requiring surgical intervention within 24 hours of diagnosis, for localized IAI infections (i.e extending beyond the organ wall but confined near the hollow viscus, mild to moderate in severity):

* Acute appendicitis: Ruptured or perforated with abscess
* Acute diverticulitis with perforation and/or abscess
* Acute cholecystitis (including gangrenous) with either rupture or perforation
* Acute gastric and duodenal ( > 24 hours) perforation
* Traumatic (> 12 hours) perforation of the intestines
* Secondary peritonitis due to perforated viscus
* Intra-abdominal abscess (including of liver and spleen)

Exclusion Criteria:

* Traumatic bowel perforation requiring surgery within 12 hours
* Perforation of gastroduodenal ulcers requiring surgery within 24 hours
* other intra-abdominal processes in which the primary etiology was unlikely to be infectious.
* Patients lactating or pregnant
* Patients with a history of allergy, hypersensitivity, or any severe reaction to the study antibiotics
* Patients with rapidly progressive or terminal illness;
* Patients with a history or presence of severe hepatic or renal disease (e.g. creatinine clearance < 0.5 ml/min/1.73 m2);
* Patients with a concomitant infection that would interfere with evaluation of response to the study antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Compare the failure rate of short therapy with Ertapenem and with AS in localized IAI | 3 days

SECONDARY OUTCOMES:
Any other complication | intraoperatively, postoperatively, at discharge, at 7-days, 1-month, 6-months follow-up
The total costs of antibiotic therapy | during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Catena, MD PhD, Study Director — S.Orsola-Malpighi University Hospital - University of Bologna; Luca Ansaloni, MD, Principal Investigator — S.Orsola-Malpighi University Hospital - University of Bologna; Giorgio Ercolani, MD, Principal Investigator — S.Orsola-Malpighi University Hospital - University of Bologna; Antonio Daniele Pinna, MD, Study Chair — S.Orsola-Malpighi University Hospital - University of Bologna; Cristina Puggioli, MD, Principal Investigator — S.Orsola-Malpighi University Hospital - University of Bologna; Salomone Di Saverio, M.D., Principal Investigator — S.Orsola-Malpighi University Hospital - University of Bologna
Locations (1):
- S.Orsola-Malpighi University Hospital - University of Bologna, Bologna, Italy

REFERENCES:
- [Background] Basoli A, Chirletti P, Cirino E, D'Ovidio NG, Doglietto GB, Giglio D, Giulini SM, Malizia A, Taffurelli M, Petrovic J, Ecari M; Italian Study Group. A prospective, double-blind, multicenter, randomized trial comparing ertapenem 3 vs >or=5 days in community-acquired intraabdominal infection. J Gastrointest Surg. 2008 Mar;12(3):592-600. doi: 10.1007/s11605-007-0277-x. Epub 2007 Sep 11. PMID 17846853
- [Derived] Catena F, Vallicelli C, Ansaloni L, Sartelli M, Di Saverio S, Schiavina R, Pasqualini E, Amaduzzi A, Coccolini F, Cucchi M, Lazzareschi D, Baiocchi GL, Pinna AD. T.E.A. Study: three-day ertapenem versus three-day Ampicillin-Sulbactam. BMC Gastroenterol. 2013 Apr 30;13:76. doi: 10.1186/1471-230X-13-76. PMID 23631512
- [Derived] Coccolini F, Catena F, Ansaloni L, Ercolani G, Di Saverio S, Gazzotti F, Lazzareschi D, Pinna AD. A prospective, multi centre, randomized clinical study to compare the efficacy and safety of Ertapenem 3 days versus Ampicillin-Sulbactam 3 days in the treatment of localized community acquired intra-abdominal infection. (T.E.A. Study: Three days Ertapenem vs three days Ampicillin-sulbactam). BMC Gastroenterol. 2011 Apr 18;11:42. doi: 10.1186/1471-230X-11-42. PMID 21501482